CLINICAL TRIAL: NCT05767840
Title: Development and Pilot Testing of an Integrated Mental Healthcare Plan for Management of Depression and Self-harm in a Rural District (Thatta) in Pakistan
Brief Title: Integrated Mental Healthcare Plan for Management of Depression and Self-harm in Pakistan
Acronym: PRIME-PK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIME-PK
Record Dates: First submitted 2023-02-28; First posted 2023-03-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Depression; Self Harm
Keywords: treatment gap; mental health; primary care; task shifting; mhGap; Pakistan
MeSH Terms: conditions — Depression; Self-Injurious Behavior; Psychological Well-Being | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mgGap-IG (Experimental): MhGap-IG intervention to be delivered to depression and self-harm cohorts
  Interventions: Other: psychological interventions

INTERVENTIONS:
Other: psychological interventions — mhGap-IG Depression and self-harm module. For participants identified as has having depression, following interventions will be offered depending on nature of the participants.
  1. Khushi Aur Khatoon - for the treatment of depression and anxiety
  2. Learning through Play Plus - 10-session group intervention that integrates parental information about child development and Cognitive Behavior Therapy
  3. Problem management Plus (PM+) - PM+ is for adults suffering from symptoms of common mental health problems , as well as self-identified practical problems.
  Cohort identified as having a recent history of self-harm will receive; Culturally Adapted Manual Assisted Problem Solving Intervention (CMAP) - This intervention is a manual-assisted intervention, adapted from a self-help guide called Life After Self-Harm.
  Other Names: mhGap-IG

SUMMARY:
Aims:

1. To describe the process of developing a feasible district mental healthcare plan (MHCP) for depression, self-harm and suicide prevention, and
2. To describe its enabling intervention packages and components to be delivered at the Basic Health Units in Thatta district.

The proposed study will be a pilot implementation with nested qualitative component. The study will also involve situational analysis for proposed study site and Theory of Change workshops with key stakeholders.

This study is a replication of the methods used in the development of a district mental healthcare plan in Uganda (Kigozi et al., 2016).

DETAILED DESCRIPTION:
Mental neurological and substance use (MNS) disorders contribute significantly to global burden of disease. The WHO Mental Health Action Programme (MhGAP) taking a life course approach has developed an intervention guide to scale up services in low and middle income countries (LMICs) focusing on priority mental health conditions in adults and older adults.

The gap between the individuals in need of mental health interventions and those who actually receive such care remains very large. To reduce the treatment gap, the WHO Mental Health Action Plan (WHO, 2017) strongly recommended assessment, diagnosis and treatment of MNS in community settings and primary healthcare (PHC). Central to this agenda is the WHO Mental Health Gap Action Programme (mhGAP) and intervention guide (IG) (WHO, 2010) which is an evidence based tool.

The proposed project aims to integrate the adapted WHO-mhGap-IG for depression, self-harm and suicide prevention into the community and primary settings in Thatta (situated in the province of Sindh, Pakistan).

Depression and self-harm are selected priority conditions for the proposed study.

In order to collect information and detailed cross-sectional data on health and factors that can influence health of Thatta district, a situational analysis tool will be used.

Both one to one in-depth interviews as well as focus groups will be conducted with stakeholders to explore possible barriers and facilitators of testing the feasibility of adapted mhGap-IG for depression and self-harm in Thatta.

Pilot study will be conducted using the mhGAP-Intervention Guide (mhGAP-IG) (two modules: Depression, self harm and suicide prevention)

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and above presenting to recruiting health facilities will be assessed by the research team for depression (positive) and/or history of self-harm (positive

Exclusion Criteria:

* Patients below 18 years of age,
* Patients taking medication for/ having a diagnosis of substance abuse, severe mental/physical disability/ comorbidity, whereby they are unable to participate in the interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Piloting log to record number of patients with depression and or self-harm episode, treatment initiated and patients referred | Recruitment From First month of study to the end of thirst month of the study start date.
  Culturally Adapted Manual Assisted Problem Solving Intervention (CMAP) - This intervention is a manual-assisted intervention which has been adapted from a self-help guide called Life After Self-Harm based on the principles of CBT

SECONDARY OUTCOMES:
Patient Health Questionnaire | Change in scores from baseline to 3rd-month follow-up on PHQ-9
  This is a10 item questionnaire with a total score ranging from 1-4 indicates minimal depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, and 20-27 severe depression. A cut-off score of 10 and above indicate high likelihood of presence of depression.
Generalised Anxiety Disorder scale | Change in scores from baseline to 3rd-month follow-up on GAD-7
  This is a 7-item scale. GAD-7 total score for the seven items ranges from 0 to 21.0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety. A cut-off score of 10 and above indicate high likelihood of presence of anxiety.
Deliberate Self-Harm Inventory | Repetition of a self-harm episode from baseline to end of 3rd month post-baseline
  DSHI will be used to collect information about episode of self-harm. is a 17-item self-report questionnaire developed to assess deliberate self-harm. It is behaviorally based and assesses aspects of deliberate self-harm such as frequency, severity, duration, and type of self-harming behavior
Oslo - 3 items social support scale | Change in scores from baseline to 3rd-month follow-up on social support
  Oslo-3 social support scale is a short three item rating scale. This scale assesses relationship with friends, family and neighbors. Each item is scored on a 5-point rating scale, and the total score ranges from 3 to 15, with high scores indicating greater level of support.
Life Events Checklist | Number of stressful events identified by each participant as present in last 12 months
  The domains that accounted for most of the life events and difficulties will be included and rated categorically as present or not in the previous 12 months.
EuroQoL-5 Dimensions | Change in scores from baseline to 3rd-month follow-up on EQ-5D
  This is a standardized instrument to measure health-related quality of life. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression)
Client Services Receipt Inventory | Change in health service utilization from baseline to 3 month follow-up recorded through CSRI
  Participants will be asked to give a detailed description of the use of health services (including the informal sector faith healers/Imams) in last 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- District health facility, Thatta, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared on request

REFERENCES:
- [Background] Kigozi FN, Kizza D, Nakku J, Ssebunnya J, Ndyanabangi S, Nakiganda B, Lund C, Patel V. Development of a district mental healthcare plan in Uganda. Br J Psychiatry. 2016 Jan;208 Suppl 56(Suppl 56):s40-6. doi: 10.1192/bjp.bp.114.153742. Epub 2015 Oct 7. PMID 26447171